CLINICAL TRIAL: NCT01527968
Title: A Prospective, Randomized, Double Blind, Double-Dummy Study Comparing the Safety and Efficacy of Epsilon Aminocaproic Acid (eACA) Versus Tranexamic Acid (TXA) Versus Placebo for Prevention of Blood Loss in Total Knee Arthroplasty
Brief Title: Epsilon Aminocaproic Acid Vs. Tranexamic Acid Vs. Placebo for Prevention of Blood Loss in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heekin Orthopedic Research Institute (Other)
Responsible Party: Principal Investigator, R. David Heekin, MD, Principal Investigator, Heekin Orthopedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 242119
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Tranexamic Acid; Aminocaproic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tranexamic Acid (Active Comparator): TXA as 10mg/kg x 1 dose in 100mL normal saline over 15 minutes prior to the procedure then an infusion of 1mg/kg/hr during the procedure + placebo (normal saline as the dummy for eACA.)
  Interventions: Drug: Tranexamic Acid
- Epsilon Aminocaproic Acid (Active Comparator): eACA as 150mg/kg in 250mL of IV normal saline over 15 minutes prior to the procedure then an infusion of 15mg/kg/hr during the procedure + placebo (normal saline as the dummy for TXA).
  Interventions: Drug: Epsilon Aminocaproic Acid
- Placebo (Placebo Comparator): Control Normal Saline x 2 infusions as the double dummy for TXA and eACA.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Tranexamic Acid — TXA as 10mg/kg x 1 dose in 100mL normal saline over 15 minutes prior to the procedure then an infusion of 1mg/kg/hr during the procedure + placebo (normal saline as the dummy for eACA.)
  Arms: Tranexamic Acid
Drug: Epsilon Aminocaproic Acid — eACA as 150mg/kg in 250mL of IV normal saline over 15 minutes prior to the procedure then an infusion of 15mg/kg/hr during the procedure + placebo (normal saline as the dummy for TXA).
  Arms: Epsilon Aminocaproic Acid
Drug: Normal Saline — Control Normal Saline x 2 infusions as the double dummy for TXA and eACA.
  Arms: Placebo

SUMMARY:
TXA and EACA have been reported to reduce blood loss in cardiac and neuro surgery, but there is no literature available comparing the two in total knee arthroplasty (TKA). The investigators want to determine if TXA or EACA compared with placebo are effective and safe for blood loss prevention in TKA by comparing blood loss, transfusion rates, and total cost.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to receive primary unilateral total knee arthroplasty

Exclusion Criteria:

* Subject requires bilateral staged total knee arthroplasty
* Religious beliefs that would limit blood transfusion
* History of acquired defective color vision (inhibits monitoring for adverse events)
* Patients with a known history of upper urinary tract bleeding
* History of abnormal coagulation
* Renal dysfunction defined by elevated BUN and CR or BUN to CR ratio of 20:1 within 30 days of surgery
* Active intravascular clotting
* Known allergy to either TXA or eACA
* Myocardial Infarct within 6 months
* History of stroke
* Patient is a prisoner

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Blood loss until the drain is removed | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: R. David Heekin, M.D., Principal Investigator — Heekin Institute for Orthopedic Research